CLINICAL TRIAL: NCT03329508
Title: A Phase 3, Twelve-week Study to Determine the Efficacy, Safety and Tolerability of P2B001 Once Daily Compared to Its Individual Components in Subjects With Early Parkinson's Disease and to a Calibration Arm of Pramipexole ER.
Brief Title: A Phase 3 Study With P2B001 in Subjects With Early Parkinson's
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharma Two B Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P2B001/003
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease; Early Parkinson's Disease
Keywords: Parkinson disease; early Parkinson's Disease; Parkinson's diagnosis; Parkinson's tretment; Parkinson's medications
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; Pramipexole

STUDY DESIGN:
Intervention Model Description: 4 arms
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- P2B001 0.6/0.75 mg (Experimental): Fixed dose combination once daily capsule of pramipexole 0.6mg and rasagiline 0.75mg, + matching placebo tablet
  Interventions: Drug: P2B001 0.6/0.75 mg
- rasagiline 0.75mg (Experimental): Rasagiline 0.75mg Once daily capsule, component of P2B001, + matching placebo tablet
  Interventions: Drug: Rasagiline 0.75 mg
- Pramipexole 0.6mg (Experimental): Pramipexole 0.6mg once daily capsule, component of P2B001 + matching placebo tablet
  Interventions: Drug: Pramipexole 0.6 mg
- Pramipexole Extended Release (Active Comparator): Marketed pramipexole ER tablet titrated to optimal dose of 1.5, 3.0 or 4.5mg + matching placebo capsule
  Interventions: Drug: Marketed Pramipexole ER

INTERVENTIONS:
Drug: P2B001 0.6/0.75 mg — Fixed low dose extended release combination capsule of pramipexole and rasagiline
  Other Names: P2B001 capsule
  Arms: P2B001 0.6/0.75 mg
Drug: Rasagiline 0.75 mg — Rasagiline 0.75 mg oral extended release capsule, component
  Other Names: RAS 0.75
  Arms: rasagiline 0.75mg
Drug: Pramipexole 0.6 mg — Pramipexole 0.6 mg oral extended release capsule, component
  Other Names: PPX 0.6
  Arms: Pramipexole 0.6mg
Drug: Marketed Pramipexole ER — Marketed Pramipexole ER titrated to optimal dose of 1.5, 3 or 4.5 mg tablet
  Other Names: PramiER
  Arms: Pramipexole Extended Release

SUMMARY:
P2B001 is an investigational drug that comprised of low doses of two drugs, pramipexole and rasagiline, which are both approved drugs and routinely used in standard therapy for Parkinson's disease. The two drugs work in two different mechanisms that help each other, so there is a reason to believe that their combined activity will be better than each individual drug, and that lower doses can be used without losing the therapeutic effect. Thus, the development of P2B001 is intended to provide a combination of low doses of these two drugs, in an improved formulation, that is hoped to be more effective in controlling Parkinson's disease symptoms and with less side effects than each of the drugs taken alone or the current available commercial drugs taken together. In a previously completed clinical trial a significant improvement in Parkinson's disease symptoms was seen in patients treated with P2B001 compared to patients that were treated with placebo.

In this phase 3 study , the safety and efficacy of P2B001 will be assessed by comparing P2B001 to its individual components pramipexole and rasagiline. This will be done by monitoring the motor and non-motor symptoms, evaluating responses participants provide on questionnaires relating to Parkinson's disease and quality of life that will be completed on every visit. In addition, this study will also compare P2B001 to a marketed drug of pramipexole ER. Approximately 525 patients will participate in this research study and the participation in this study will last between 14 to 18 weeks.

DETAILED DESCRIPTION:
A total of 525 eligible subjects with early untreated Parkinson's disease (PD), will be randomized to 4 treatment groups. Each subject will participate in the study for approximately 18 weeks including a 30 day screening period, 12 week treatment period, and 2 weeks follow-up period. Subjects will be requested to take one capsule and 1-3 tablets of study drug by mouth with a glass of water every day for 13 weeks. The study requires seven visits to the clinic one every 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Parkinson's disease consistent with the UK Brain Bank Criteria and must have bradykinesia with sequence effect. If rest tremor does not exist must have prominent asymmetry of motor function.
2. Subject with disease duration less than 3 years since diagnosis.
3. Subject has a H&Y stage score of < 3.
4. Subject has a MMSE score ≥ 26.

Exclusion Criteria:

1. Subject has an atypical parkinsonian syndrome or secondary parkinsonism
2. Subject has previous exposure to levodopa or a dopamine agonist for longer than 4 weeks; if previous exposure was less than 4 weeks then it must not be within 2 months prior to the baseline visit.
3. Subject has previous exposure to a MAO-B inhibitor for longer than 4 weeks; if previous exposure was less than 4 weeks then it must not be within 3 months prior to the baseline visit.
4. Subject who has taken anticholinergic drugs for PD or amantadine for longer than 4 weeks; if previous exposure was less than 4 weeks then it must not be within 1 month prior to the baseline visit.
5. Subject has moderate (Child-Pugh categorization B, score 7-9) or severe (Child-Pugh categorization C, score 10-15) hepatic impairment.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pninit Litman, Study Director — Pharma2b LTD
Locations (71):
- United States (45):
  - P2B001/003 Site Scottsdale, Scottsdale, Arizona
  - P2B001/003 study site Scottsdale, Scottsdale, Arizona
  - P2B001/003 Study site little Rock, Little Rock, Arkansas
  - P2B001 site Los Angeles, Los Angeles, California
  - P2B001 Study site Englewood,, Englewood, Colorado
  - P2B001 Study Vernon, Vernon, Connecticut
  - P2B001/003 site Boca Raton, Boca Raton, Florida
  - P2B001/003 Site Boca Raton, Boca Raton, Florida
  - P2B001/003 study site Jacksonville, Jacksonville, Florida
  - P2B001/003 site Miami, Miami, Florida
  - P2B001/003 Site Port Charlotte, Port Charlotte, Florida
  - P2B001/003 Site Sarasota, Sarasota, Florida
  - P2B001/003 Site Tampa, Tampa, Florida
  - P2B001/003 Site Augusta, Augusta, Georgia
  - P2B001/003 study site Honolulu, Honolulu, Hawaii
  - P2B001/003 site Chicago, Chicago, Illinois
  - P2B001/003 Site Winfield, Winfield, Illinois
  - P2B001/003 site Kansas City, Kansas City, Kansas
  - P2B001/003 Site Lexington, Lexington, Kentucky
  - P2B001/003 study site Boston, Boston, Massachusetts
  - P2B001/003 Site East Lansing, East Lansing, Michigan
  - P2B001/003 study site west Bloomfield, West Bloomfield, Michigan
  - P2B001/003 Site Golden Valley, Golden Valley, Minnesota
  - P2B001/003 site St. Louis, St Louis, Missouri
  - P2B001/003 study site New Hampshire, Lebanon, New Hampshire
  - P2B001/003 Study site Camden, Camden, New Jersey
  - P2B001 Study site Edison, Edison, New Jersey
  - P2B001/003 Study site Albuquerque, Albuquerque, New Mexico
  - P2B001/003 Study site Brooklyn, Brooklyn, New York
  - P2B001/003 Site Commack, Commack, New York
  - P2B001/003 New York, New York, New York
  - P2B001 Study site Syracuse, Syracuse, New York
  - P2B001/003 Study site Williamsville, Williamsville, New York
  - P2B001/003 Site Asheville, Asheville, North Carolina
  - P2B001 study site Cincinnati, Cincinnati, Ohio
  - P2B001/003 Site Toledo, Toledo, Ohio
  - P2B001/003 Study site Hershey, Hershey, Pennsylvania
  - P2B001/003 Greenville, Greenville, South Carolina
  - P2B0011/003 Study Veracity Neuroscience, Memphis, Tennessee
  - p2B001/003 Study site Memphis, Memphis, Tennessee
  - P2B001/003 Study site Nashville, Nashville, Tennessee
  - P2B001/003 Site Dallas, Dallas, Texas
  - P2B001/003 Study site Alexandria, Alexandria, Virginia
  - P2B001/003, Falls Church, Virginia
  - P2B001/003 Site Kirkland, Kirkland, Washington
- P2B001/003 study site Toronto, Toronto, Ontario, Canada
- Germany (14):
  - P2B001/003 Study site Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - P2B001/003 study site Ulm, Ulm, Baden-Wurttemberg
  - P2B001/003 study site Haag, Haag, Bavaria
  - P2B001/003 Study site Haag, Haag, Bavaria
  - P2B001/003 Study site München, München, Bavaria
  - P2B001/003 Study site Hanau, Hanau, Hesse
  - P2B001/003 Study site Bochum, Bochum, North Rhine-Westphalia
  - P2B001/003 Study site Münster, Münster, North Rhine-Westphalia
  - P2B001/003 Study site Dresden, Dresden, SaACHSEN
  - P2B001/003 study site Leipzig, Leipzig, Saxony
  - P2B001/003 study site Gera Germany, Gera, Thuringia
  - P2B001/003 Study site Gera, Gera, Thuringia
  - P2B001/003 Study site Berlin, Berlin
  - P2B001/003 site Munich, Munich
- Spain (11):
  - P2B001/003 Study site Sant Cugat del Vallés, Sant Cugat Del Vallés, Barcelona
  - P2B001/003 study site Mostoles, Móstoles, Madridid
  - P2B001/003 Study site Pamplona, Pamplona, Navarre
  - P2B001/003 Study site La Paz, Madrid, S
  - P2B001/003 Study site Barcelona, Barcelona
  - P2B001/003 Study site Vall d'Hebrón, Barcelona
  - P2B001/003 Study site Navarra Madrid, Madrid
  - P2B001/003 study site Madrid, Madrid
  - P2B001/003 Study site Madrid, Madrid
  - P2B0011/003 Study site HM Centro Integral de Neurociencias (CINAC), Madrid
  - P2B001/003 Study site Puerta de Hierro - Majadahonda, Majadahonda

RESULTS

PARTICIPANT FLOW:
Groups:
- P2B001: Fixed dose combination once daily capsule of pramipexole and rasagiline
  P2B001: Fixed dose once daily combination capsule of pramipexole and rasagiline
- Rasagiline Capsule: rasagiline Once daily capsule
  Rasagiline: Rasagiline oral capsule
- Pramipexole Capsule: Pramipexole once daily capsule
  Pramipexole: Pramipexole low dose oral capsule
- Pramipexole Extended Release: pramipexole ER tablet titrated to optimal dose of 1.5, 3.0 or 4.5mg
  Pramipexole ER: Pramipexole ER titrated to optimal dose
Period: Overall Study
Arm/Group | P2B001 | Rasagiline Capsule | Pramipexole Capsule | Pramipexole Extended Release
Started | 157 | 154 | 156 | 77
Completed | 137 | 134 | 137 | 67
Not Completed | 20 | 20 | 19 | 10

BASELINE CHARACTERISTICS:
Population: The dispensing of the investigational product was based on a "just-in-time" shipping strategy per subject. Randomization was done at the end of the Screening period and before the Baseline Visit to allow for shipping of the kit to the site. Twenty-five (25) subjects were enrolled and randomized into treatment groups, but withdrew from study prior to first dose. They did not came to baseline visit , receive study drug nor did they receive a post-randomization evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | P2B001 | Rasagiline Capsule | Pramipexole Capsule | Pramipexole Extended Release | Total
Number analyzed (Participants) | 157 | 154 | 156 | 77 | 544
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 79 | 71 | 77 | 41 | 268
  >=65 years | 78 | 83 | 79 | 36 | 276
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (9) | 65 (1) | 64 (9) | 63 (9) | 64 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 52 | 24 | 175
  Male | 106 | 106 | 104 | 53 | 369
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 3
  Asian | 0 | 3 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 2 | 0 | 5
  Black or African American | 2 | 3 | 5 | 1 | 11
  White | 150 | 145 | 147 | 74 | 516
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 0 | 1 | 0 | 2
  United States | 109 | 109 | 108 | 54 | 380
  Germany | 29 | 29 | 30 | 15 | 103
  Spain | 18 | 16 | 17 | 8 | 59
Total UPDRS [Mean (Standard Deviation); unit: units on a scale] — Unified Parkinson's Disease Rating Scale , score 0-160 minimum is 0 and maximum is 160 points . High score mean worse outcome Population: Twenty-five (25) subjects as explained above were enrolled and randomized into treatment groups, but withdrew from study prior to first dose. They did not came to baseline visit , receive study drug nor did they receive a post-randomization evaluation. The baseline was measured to 519 subjects who came to baseline visit , had assessment and took at least one dose of study medication . These are also the safety dataset.
  units on a scale
    number analyzed (Participants) | 150 | 148 | 147 | 74 | 519
    (all) | 30.7 (9.9) | 31.3 (10.2) | 31.3 (11.0) | 28.8 (10.0) | 30.8 (10.3)
Epworth Sleepiness Score [Mean (Standard Deviation); unit: units on a scale] — scale from 0-24. Minimum is 0 and maximum 24. high score mean worse outcome Population: Twenty-five (25) subjects as explained above were enrolled and randomized into treatment groups, but withdrew from study prior to first dose. They did not came to baseline visit , receive study drug nor did they receive a post-randomization evaluation. The baseline was measured to 519 subjects who came to baseline visit , had assessment and took at least one dose of study medication . These are also the safety dataset.
  units on a scale
    number analyzed (Participants) | 150 | 147 | 148 | 74 | 519
    (all) | 5.5 (4.0) | 5.7 (4.3) | 6.2 (4.0) | 6.1 (4.1) | 5.8 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Unified Parkinson's Disease Rating Scale (UPDRS) Score (Defined as Sum of Parts II and III, Scores (0-160).
Description: Differences between P2B 0.6/0.75 mg as compared to its individual components in the change of total UPDRS score (defined as sum of parts II and III, scores (0-160).
  UPDRS- Unified Parkinson's Disease Rating Scale, minimum value is 0 points and maximum value is 160.
  High score mean worse outcome.
Time Frame: baseline to week 12
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | P2B001 | Rasagiline Capsule | Pramipexole Capsule | Pramipexole Extended Release
Number analyzed (Participants) | 147 | 144 | 144 | 72
score on a scale | -7.98 (0.60) | -4.69 (0.61) | -5.32 (0.61) | -8.35 (0.86)
Statistical Analysis 1: Comparison: P2B001 vs Pramipexole Capsule; Test type: Superiority; p = 0.0018, MMRM; Differences of Least Square Means = -2.66, 95% CI 2-sided [-4.33 to -1.0], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: P2B001 vs Rasagiline Capsule; Test type: Superiority; p = 0.0001, MMRM; Mean Difference (Net) = -3.30, 95% CI 2-sided [-4.96 to -1.63], Standard Error of Mean 0.85

2. Secondary Outcome: Change in Epworth Sleepiness Scale (ESS) Score.
Description: Differences between P2B 0.6/0.75 mg as compared to pramipexole ER tablets in the change of Epworth Sleepiness Scale (ESS) score.
  Scale is 0-24 , when 24 is worse outcome
Time Frame: baseline to week 12
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | P2B001 | Rasagiline Capsule | Pramipexole Capsule | Pramipexole Extended Release
Number analyzed (Participants) | 147 | 144 | 144 | 72
score on a scale | -0.33 (0.25) | -0.81 (0.26) | 0.39 (0.25) | 2.33 (0.36)
Statistical Analysis 1: Comparison: P2B001 vs Pramipexole Extended Release; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Net) = -2.66, 95% CI 2-sided [-3.50 to -1.81], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: P2B001 vs Pramipexole Extended Release; Test type: Superiority; p < 0.05, MMRM; Mean Difference (Final Values) = -2.66, 95% CI 2-sided [-3.50 to -1.81], Standard Error of Mean 0.43

3. Secondary Outcome: Change From Baseline to Week 12 in Total UPDRS III Motor
Description: Differences between P2B 0.6/0.75 mg as compared to its individual components in the change of Motor UPDRS score (UPDRS Part III ).
  UPDRS- Unified Parkinson's Disease Rating Scale, part III motor . min is 0 and Max is 108 (Worse outcome)
Time Frame: baseline to week 12
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | P2B001 | Rasagiline Capsule | Pramipexole Capsule | Pramipexole Extended Release
Number analyzed (Participants) | 147 | 144 | 144 | 72
score on a scale | -5.82 (0.47) | -4.07 (0.48) | -4.30 (0.48) | -6.36 (0.68)
Statistical Analysis 1: Comparison: P2B001 vs Pramipexole Capsule; Test type: Superiority; p = 0.0231, MMRM; Mean Difference (Net) = -1.52, 95% CI 2-sided [-2.84 to -0.21], Standard Error of Mean 0.67
Statistical Analysis 2: Comparison: P2B001 vs Rasagiline Capsule; Test type: Superiority; p = 0.0092, MMRM; Mean Difference (Net) = -1.75, 95% CI 2-sided [-3.06 to -0.43], Standard Error of Mean 0.67

4. Secondary Outcome: Change From Baseline to Week 12 in Total UPDRS II ADL
Description: Differences between of P2B 0.6/0.75 mg as compared to its individual components in the change of ADL UPDRS score (UPDRS part II) Activity of daily Life UPDRS part II minimum is 0 point and max is 52 point (worse outcome)
Time Frame: Baseline to week 12
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | P2B001 | Rasagiline Capsule | Pramipexole Capsule | Pramipexole Extended Release
Number analyzed (Participants) | 147 | 144 | 144 | 72
score on a scale | -2.14 (0.22) | -0.62 (0.22) | -0.97 (0.22) | -2.02 (0.31)
Statistical Analysis 1: Comparison: P2B001 vs Pramipexole Capsule; Test type: Superiority; p = 0.0001, MMRM; Mean Difference (Net) = -1.17, 95% CI 2-sided [-1.77 to -0.57], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: P2B001 vs Rasagiline Capsule; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Net) = -1.52, 95% CI 2-sided [-2.13 to -0.92], Standard Error of Mean 0.31

5. Secondary Outcome: Change From Baseline to End of Week 12 Visit in ADL Subscale of PDQ39
Description: The efficacy of P2B 0.6/0.75 mg as compared to Pramipexole ER tablet titrated to optimal dose.
  ADL PDQ39- Activity of daily life part in Parkinson's Disease Questionaries' 39 Score 0-100 when 100 is the worse outcome
Time Frame: Baseline to week 12
Population: mITT
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | P2B001 | Rasagiline Capsule | Pramipexole Capsule | Pramipexole Extended Release
Number analyzed (Participants) | 147 | 144 | 144 | 72
score on a scale | -5.30 (0.89) | -2.04 (0.92) | -3.40 (0.90) | -3.12 (1.27)
Statistical Analysis 1: Comparison: P2B001 vs Pramipexole Extended Release; Test type: Superiority; p = 0.1589, MMRM; Mean Difference (Net) = -2.18, 95% CI 2-sided [-5.21 to 0.85], Standard Error of Mean 1.54

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | P2B001 | Rasagiline Capsule | Pramipexole Capsule | Pramipexole Extended Release
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/147 | 0/148 | 0/74
Serious Adverse Events (participants affected / at risk) | 3/150 | 2/147 | 3/148 | 0/74
Other Adverse Events (participants affected / at risk) | 78/150 | 52/147 | 86/148 | 54/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P2B001 (N=150) | Rasagiline Capsule (N=147) | Pramipexole Capsule (N=148) | Pramipexole Extended Release (N=74)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 (2) | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
corona virus (Infections and infestations) | 0 | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P2B001 (N=150) | Rasagiline Capsule (N=147) | Pramipexole Capsule (N=148) | Pramipexole Extended Release (N=74)
nausea (Gastrointestinal disorders) | 28 (33) | 10 (10) | 24 (29) | 17 (22)
fatigue (General disorders) | 23 (27) | 2 (2) | 22 (25) | 13 (14)
somnolence (Nervous system disorders) | 22 (25) | 7 (7) | 27 (32) | 23 (29)
dizziness (Nervous system disorders) | 16 (18) | 19 (21) | 14 (15) | 7 (7)
insomnia (Psychiatric disorders) | 13 (14) | 4 (4) | 9 (9) | 7 (8)
headache (Nervous system disorders) | 9 (14) | 9 (12) | 14 (15) | 5 (5)
constipation (Gastrointestinal disorders) | 6 (6) | 9 (9) | 11 (12) | 7 (7)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 10 (11) | 4 (4)
fall (Injury, poisoning and procedural complications) | 6 (6) | 5 (12) | 8 (10) | 1 (2)
memory impairment (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 4 (4) | 5 (6) | 9 (9)
Decreased appetite (Gastrointestinal disorders) | 3 (4) | 2 (3) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03329508/Prot_000.pdf
  • Statistical Analysis Plan: SAP P2B protocol P2B001_003 NCT03329508 2021_10_21 (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT03329508/SAP_001.pdf
  • Statistical Analysis Plan: Addendum to Statistical Analysis (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT03329508/SAP_002.pdf
  • Informed Consent Form (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03329508/ICF_003.pdf